CLINICAL TRIAL: NCT01010503
Title: Evaluation of Adherence and Persistence to Tocilizumab in Combination With Methotrexate or Tocilizumab Monotherapy in Patients With Moderate to Severe Active Rheumatoid Arthritis in Local Environment.
Brief Title: A Study of Tocilizumab With or Without Methotrexate in Patients With Rheumatoid Arthritis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22508; 2009-011520-53
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — tocilizumab 8 mg/kg intravenous infusion once in 4 weeks

SUMMARY:
This open-label, single-arm, non-randomized study will evaluate the adherence and persistence to tocilizumab therapy in patients with moderate to severe active rheumatoid arthritis, who have an inadequate clinical response to non-biologic DMARDs. Patients will receive tocilizumab 8 mg/kg as intravenous infusion once every 4 weeks in combination with methotrexate or in case of intolerance to methotrexate as monotherapy. The anticipated time of study treatment is 6 months. The target sample size is 20-50 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >/= 18 years of age
* moderate to severe active rheumatoid arthritis
* inadequate response, or intolerance to previous therapy with one or more traditional DMARDs
* DAS >3.6
* pneumology examination (including chest x-ray and quantiferon)

Exclusion Criteria:

* < 18 years of age
* active infection
* active tuberculosis
* uncontrolled hyperlipoproteinaemia
* demyelinating disorders
* concomitant anti-TNF drugs
* history of intestinal ulceration and diverticulitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Piešťany, Slovakia

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 Milligrams Per Kilogram (mg/kg): Participants received tocilizumab 8 mg/kg intravenously (IV) once every 4 weeks for a maximum of 20 weeks (total of 6 infusions).
Period: Overall Study
Arm/Group | Tocilizumab 8 Milligrams Per Kilogram (mg/kg)
Started | 32
Completed | 30
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg IV once every 4 weeks for a maximum of 20 weeks (total of 6 infusions).
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.38 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Slovakia | 32
Disease Duration [Mean (Standard Deviation); unit: years] | 11.97 (10.55)
Disease Phase/Stage [Number; unit: participants] — Disease stages/phases of rheumatoid arthritis (RA): Stage I represents synovitis: synovial membrane becomes hyperemic and edematous; joint effusions with high cell count; x-rays will as yet show no destructive changes, but soft tissue swelling or osteoporosis may be seen; Stage II: inflamed synovial tissue now proliferates and begins to grow into joint cavity across articular cartilage, which it gradually destroys; Stage III: pannus of synovium; eroded articular cartilage and exposed subchondral bone x-rays will show extensive cartilage loss; Stage IV represents end-stage disease.
  participants
    Phase/Stage I | 4
    Phase/Stage II | 12
    Phase/Stage III | 12
    Phase/Stage IV | 4
Functional Class of Disease [Number; unit: participants] — Classification of global functional status in RA is as follows: Class I: completely able to perform usual activities of daily living (self-care, vocational, and avocational); Class II: able to perform usual self-care and vocational activities, but limited in avocational activities; Class III: able to perform usual self-care activities, but limited in vocational and avocational activities; and Class IV: limited in ability to perform usual self-care, vocational, and avocational activities.
  participants
    Class I | 0
    Class II | 10
    Class III | 22
    Class IV | 0
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/L] — CRP was measured in milligrams per liter (mg/L)
  mg/L | 17.84 (21.30)
Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: mm/hr] — ESR was measured in millimeters per hour (mm/hr)
  mm/hr | 55.81 (25.05)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Adherent to Original Treatment
Description: Adherence rate to original treatment according to the protocol included all participants that received the study drug beginning from Week 8 and remaining until the end of the study. This number represents participants with no changes in treatment protocol, participants with treatment discontinuation, and participants with dose reduction, but not participants that withdrew from the study prematurely.
Time Frame: Week 24
Population: Intent-to-treat population (ITT), all enrolled participants who received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
percentage of participants | 93.75

2. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28)
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) and Patient's Global Assessment of Disease Activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 ≤3.2 equals (=) low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Weeks 0, 4, 12, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
units on a scale
  Week 0 (n=32) | 7.02 (0.66)
  Week 4 (n=32) | 4.30 (1.04)
  Week 12 (n=30) | 2.85 (1.11)
  Week 24 (n=30) | 2.57 (0.91)

3. Primary Outcome: Percentage of Participants Receiving Less Than or Equal to (≤) 1 Dose of Study Drug Who Discontinued Treatment for Any Reason
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
percentage of participants | 3.13

4. Primary Outcome: Percentage of Participants Receiving Greater Than (>) 1 Dose Who Discontinued Treatment for Any Reason
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
percentage of participants | 0

5. Primary Outcome: Percentage of Participants Withdrawing From the Study Prematurely for Any Reason
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
percentage of participants | 6.25

6. Primary Outcome: Percentage of Participants With Dose Reduction to Tocilizumab 4 mg/kg
Time Frame: Weeks 0, 4, 8, 12, 16, and 20
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
percentage of participants | 18.75

7. Secondary Outcome: Patient Global Assessment of Pain
Description: Participants were asked to rate their pain using a 0 to 100 mm visual analog scale (VAS), where 0 mm = no pain and 100 mm = worst possible pain. The participant was asked to mark the line corresponding to their perceived level of pain and the distance in mm from the left edge of the scale was measured.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
units on a scale
  Week 0 (n=32) | 59.91 (14.66)
  Week 4 (n=32) | 36.31 (17.10)
  Week 8 (n=30) | 22.3 (15.79)
  Week 12 (n=30) | 17.30 (14.00)
  Week 16 (n=30) | 18.93 (14.59)
  Week 20 (n=30) | 16.73 (15.11)
  Week 24 (n=30) | 14.87 (11.32)

8. Secondary Outcome: Patient Global Assessment of Disease Activity
Description: The participant's assessment of disease activity was performed using a 100 mm VAS ranging from no activity (0) to maximal activity (100). The participant was asked to mark the line corresponding to their perceived level of disease activity and the distance in mm from the left edge of the scale was measured.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
units on a scale
  Week 0 (n=32) | 61.75 (11.76)
  Week 4 (n=32) | 35.59 (16.62)
  Week 8 (n=30) | 22.20 (14.86)
  Week 12 (n=30) | 18.20 (14.57)
  Week 16 (n=30) | 18.80 (13.42)
  Week 20 (n=30) | 18.13 (18.49)
  Week 24 (n=30) | 15.47 (12.62)

9. Secondary Outcome: Physician's Global Assessment of Disease Activity
Description: Physician's global assessment of disease activity was performed using a 100 mm VAS ranging from no arthritis activity (0) to maximal arthritis activity (100). The physician was asked to mark the line corresponding to their perceived level of the participant's disease activity and the distance in mm from the left edge of the scale was measured.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
units on a scale
  Week 0 (n=32) | 59.63 (7.89)
  Week 4 (n=32) | 27.75 (14.00)
  Week 8 (n=30) | 17.40 (9.96)
  Week 12 (n=30) | 14.20 (9.93)
  Week 16 (n=30) | 13.00 (8.68)
  Week 20 (n=30) | 12.77 (10.17)
  Week 24 (n=30) | 12.47 (8.22)

10. Secondary Outcome: Swollen Joint Count (SJC)
Description: The following 28 joints were assessed by the physician for swelling: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2). Joints were rated as 0=not swollen or 1=swollen. The total number was calculated from all the joints for a maximum score of 28.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
swollen joints
  Week 0 (n=32) | 26.66 (7.11)
  Week 4 (n=32) | 12.03 (8.24)
  Week 8 (n=30) | 7.00 (6.52)
  Week 12 (n=30) | 5.33 (6.47)
  Week 16 (n=30) | 5.33 (6.33)
  Week 20 (n=30) | 4.20 (5.088)
  Week 24 (n=30) | 4.00 (5.24)

11. Secondary Outcome: Tender Joint Count (TJC)
Description: The following 28 joints were assessed by the physician for tenderness: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2). Joints were rated as 0=not tender or 1=tender. The total number was calculated from all the joints for a maximum score of 28.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
tender joints
  Week 0 (n=32) | 16.16 (5.18)
  Week 4 (n=32) | 5.53 (5.16)
  Week 8 (n=30) | 1.97 (2.01)
  Week 12 (n=30) | 1.30 (1.68)
  Week 16 (n=30) | 1.00 (1.20)
  Week 20 (n=30) | 0.83 (1.315)
  Week 24 (n=30) | 0.63 (1.00)

12. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR indirectly measures how much inflammation is in the body. A higher ESR is indicative of increased inflammation.
Time Frame: Weeks 0, 4, 12, 20, and 24
Population: TT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
mm/hr
  Week 0 (n=32) | 55.81 (25.05)
  Week 4 (n=32) | 16.69 (10.88)
  Week 12 (n=30) | 15.23 (14.78)
  Week 20 (n=30) | 14.17 (17.81)
  Week 24 (n=30) | 11.00 (7.94)

13. Secondary Outcome: C-Reactive Protein (CRP)
Description: CRP is an acute phase protein. Levels of CRP increase with inflammation.
Time Frame: Weeks 0, 4, 12, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
mg/L
  Week 0 (n=32) | 17.84 (21.30)
  Week 4 (n=32) | 5.03 (6.07)
  Week 12 (n=30) | 5.54 (9.22)
  Week 20 (n=30) | 6.71 (13.9)
  Week 24 (n=30) | 2.97 (0.70)

14. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) Score
Description: The HAQ-DI was used to assess the physical ability and functional status of participants as well as quality of life. The disability dimension consists of 20 multiple choice items concerning difficulty in performing 8 common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Participants choose from 4 response categories, ranging from 'without any difficulty' (Score=0) to 'unable to do' (Score=3). The overall score is the average of each of the 8 category scores and ranges from 0 to 3, where 0 represents no disability and 3 very severe, high-dependency disability.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
scores on a scale
  Week 0 (n=32) | 1.77 (0.43)
  Week 4 (n=32) | 1.56 (0.49)
  Week 8 (n=30) | 1.31 (0.65)
  Week 12 (n=30) | 1.28 (0.65)
  Week 16 (n=30) | 1.23 (0.64)
  Week 20 (n=30) | 1.20 (0.644)
  Week 24 (n=30) | 1.16 (0.63)

15. Secondary Outcome: Short Form-36 (SF-36)
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 8 subscales (physical function, pain, general and mental health, vitality, social function, physical and emotional health) which can be aggregated to derive a physical-component summary score and a mental-component summary score. Scores for each subscale range from 0 to 10, and the composite scores range from 0 to 100, with higher scores indicating better health.
Time Frame: Weeks 0, 12, and 24
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32
scores on a scale
  Physical Functioning, Week 0 (n=32) | 26.08 (18.09)
  Physical Functioning, Week 12 (n=30) | 44.50 (27.58)
  Physical Functioning, Week 24 (n=30) | 47.22 (31.92)
  Role limits due to physical health, Week 0 (n=32) | 6.25 (18.71)
  Role limits due to physical health, Week 12 (n=30) | 49.17 (45.34)
  Role limits due to physical health, Week 24 (n=30) | 44.44 (45.60)
  Role limits due to emotional prob., Week 0 (n=32) | 16.67 (34.23)
  Role limits due to emotional prob., Week 12 (n=30) | 61.11 (45.34)
  Role limits due to emotional prob., Week 24 (n=30) | 55.56 (48.47)
  Energy/fatigue, Week 0 (n=32) | 30.31 (17.93)
  Energy/ fatigue, Week 12 (n=30) | 48.33 (26.14)
  Energy/fatigue, Week 24 (n=30) | 50.00 (31.32)
  Emotional well-being, Week 0 (n=32) | 50.00 (19.10)
  Emotional well-being, Week 12 (n=30) | 63.70 (24.16)
  Emotional well-being, Week 24 (n=30) | 65.33 (32.92)
  Social functioning, Week 0 (n=32) | 39.45 (17.61)
  Social functioning, Week 12 (n=30) | 60.83 (25.36)
  Social functioning, Week 24 (n=30) | 62.50 (35.11)
  Pain, Week 0 (n=32) | 28.67 (15.34)
  Pain, Week 12 (n=30) | 55.75 (27.63)
  Pain, Week 24 (n=30) | 56.11 (33.32)
  General health, Week 0 (n=32) | 38.28 (10.82)
  General health, Week 12 (n=30) | 46.83 (16.32)
  General health, Week 24 (n=30) | 46.25 (23.41)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) related to study medication were reported irrespective of elapsed time from last administration of study medication. Non-related SAEs were reported during the study period and 28 days after the last dose of study medication.
Arm/Group | Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 10/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=32)
Crash of left foot local infection of skin and subcutaneous tissue (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Lumbago (Musculoskeletal and connective tissue disorders) | 1
Congestive heart failure (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab 8 mg/kg (N=32)
Hepatopathy (Hepatobiliary disorders) | 2 (2)
Leucopenia+lymphopenia (Blood and lymphatic system disorders) | 3 (3)
Acute bronchitis (Reproductive system and breast disorders) | 3 (3)
Acute nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute pulpitis (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights